CLINICAL TRIAL: NCT03473808
Title: Brain Functional Connectivity & Sensory Stimulation-enhanced Therapy Post Stroke
Brief Title: Functional Connectivity & Stimulation-enhanced Therapy Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); University of Delaware (Other)
Responsible Party: Principal Investigator, Na Jin Seo, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO74041; U54GM104941 (NIH)
Record Dates: First submitted 2018-03-05; First posted 2018-03-22 (Actual); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Stroke
Keywords: Hand Function; Occupational Therapy; Physical Stimulation
MeSH Terms: conditions — Stroke | interventions — Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- therapy + vibration (Experimental): Imperceptible vibration applied to the wrist during a standardized hand task practice therapy program.
  Interventions: Behavioral: task-practice therapy; Other: Vibration

INTERVENTIONS:
Behavioral: task-practice therapy — Standardized hand therapy program
Other: Vibration — Peripheral vibration applied to the wrist skin at an imperceptible level

SUMMARY:
After stroke, it is common for individuals to experience hand impairment. This deficit can severely restrict functional ability and independence. Recovery of hand function following stroke is highly variable. In this study, the investigators will use brain imaging to predict individual response to treatment. Survivors of stroke will receive upper extremity therapy while they concurrently receive imperceptible vibration to the wrist aimed to enhance therapy outcomes.

DETAILED DESCRIPTION:
The ability to predict individuals' responses to treatment can enable effective allocation of a treatment to likely responders. The long-term goal is to determine whether acute changes in brain functional connectivity immediately after one treatment session can predict ultimate gains in motor function after completing multiple treatment sessions. The objective of this study is to determine feasibility and to examine association between change in brain functional connectivity after one session and motor gains after completion of all treatment sessions. This study is a prospective single-cohort longitudinal study. The treatment is task-practice therapy (3d/wk, 18-session) accompanied with concurrent imperceptible wrist vibration that is intended to prime the cortical sensorimotor network and enhance hand functional recovery in chronic stroke survivors. Hand function will be assessed before/after therapy and at 1-month follow-up. Connectivity will be assessed using fMRI and EEG before and after a treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 or older
* At least 6 months post-stroke
* Moderate upper limb impairment with the ability to participate in hand task practices
* Fingertip touch sensory deficits (e.g., Monofilament>2.83, 2-point discrimination>5mm, sense of numbness, tingling)

Exclusion Criteria:

* Complete upper limb deafferentation
* Rigidity (Modified Ashworth Scale=5)
* Botulinum toxin injection within 3 months prior to enrollment or during enrollment
* Brainstem stroke
* Comorbidity (peripheral neuropathy, orthopaedic conditions in the hand that limit ranges of motion, premorbid neurologic conditions, compromised skin integrity of the hand/wrist due to long-term use of blood thinners)
* Concurrent upper extremity rehabilitation therapy
* Language barrier or cognitive impairment that precludes following instructions or providing consent
* MRI incompatible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Kautz, PhD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapy + Vibration
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Therapy + Vibration
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (5.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hand Motor Function
Description: Change in hand motor function as measured by the Box and Block Test. The test measures the number of blocks that a participant moves within one minute. The scale ranges from 0 to a positive number. Higher numbers represent better outcomes.
Time Frame: Baseline to approximately 1 week after the completion of 18 therapy sessions.
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | Therapy + Vibration
Number analyzed (Participants) | 4
blocks | 0.83 (3.09)

2. Primary Outcome: Mean Change in Hand Motor Function
Description: as for outcome 1
Time Frame: Baseline to approximately 4 weeks after the completion of 18 therapy sessions.
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | Therapy + Vibration
Number analyzed (Participants) | 4
blocks | 0.21 (1.18)

3. Secondary Outcome: Mean Change in Hand Motor Function
Description: Change in hand motor function as measured by the Wolf Motor Function Test Time. This test measures time to complete upper extremity movements in seconds. More negative values represent a greater reduction in time, thus better outcomes.
Time Frame: Baseline to approximately 1 week after the completion of 18 therapy sessions.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Therapy + Vibration
Number analyzed (Participants) | 4
seconds | -10.09 (3.66)

4. Secondary Outcome: Mean Change in Hand Motor Function
Description: as for outcome 3
Time Frame: Baseline to approximately 4 weeks after the completion of 18 therapy sessions.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Therapy + Vibration
Number analyzed (Participants) | 4
seconds | -14.24 (5.51)

ADVERSE EVENTS:
Time Frame: Baseline through one month follow-up (10 weeks).
Arm/Group | Therapy + Vibration
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy + Vibration (N=5)
Root Canal (Surgical and medical procedures) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (General disorders) | 1 (2)
Temporary increase in muscle tone (Musculoskeletal and connective tissue disorders) | 1 (3)
Bumped affected upper extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Temporary upper extremity numbness (Nervous system disorders) | 2 (2)
Temporary skin irritation (Skin and subcutaneous tissue disorders) | 2 (7)
Worsening Monofilament Score (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT03473808/Prot_SAP_000.pdf